CLINICAL TRIAL: NCT05863338
Title: The Effect of Nursing Follow-Up by Phone on the Self-Efficacy, Pain and Disease Activity Level of Individuals Diagnosed With Rheumatoid Arthritis Using Biological Agents
Brief Title: The Effect of Nursing Follow-Up by Phone on The Self-Efficacy,Pain,Disease Activity in Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Done Gunay, PhD student, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-06/38
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Tele-nursing
Keywords: Rheumatoid Arthritis; Biological Agent; Telephone Monitoring; Nursing Practices
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: The study was conducted as the randomized controlled experimental trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Data collection tools were applied face to face. Patient education was carried out in the polyclinic. A training booklet was given at the end of the training. Afterwards, patients were called once a week by telephone for 12 weeks. The patients were followed up by the nurse over the phone and counseling was provided to the patients. Patients were able to call the research nurse when needed. Interim evaluation was made at the 12th week. Data collection tools were applied face-to-face in the outpatient clinic. Patients 13-24. Between weeks, 12 more phone calls were made, once a week. The patients were followed up by the nurse by telephone, and the patients continued to receive counseling services. Patients were able to call the research nurse when needed. At the end of the 24th week, the research forms were applied face to face in the outpatient clinic. The research has finished.
  Interventions: Behavioral: NURSING FOLLOW-UP BY PHONE
- Control Group (No Intervention): Individuals meeting the sample specifications were included in the control group in accordance with the order of numbers in the lists created by randomly assigning numbers. Data collection tools were applied face to face. Routine outpatient follow-ups continued. Interim evaluation was made at the 12th week. In the interim evaluation, data collection tools were applied face to face. Then, routine outpatient follow-up between 13 and 24 weeks continued. At the end of the 24th week, data collection tools were applied face to face. The patients were educated in the outpatient clinic. A training booklet was given at the end of the training. The research has been terminated.

INTERVENTIONS:
Behavioral: NURSING FOLLOW-UP BY PHONE — The training was carried out in the form of individual training and as a single session.The training,which lasted about 30 minutes,was carried out in the training room of the polyclinic with the support of Barco vision.In the training session,lecture,question-answer methods were used and at the end of the training session,a booklet containing the training content was given to the patients.The researcher phoned the patients once a week for 24 weeks,conveyed how they were doing,whether there was anything they wanted to ask or learn,and provided counseling to the patients in line with their needs.The next week's plan was also determined in the phone calls made in the following weeks.Patient follow-ups as stated were continued for 24 weeks.At the 12th and 24th weeks of the telephone nursing follow-up, the patients filled out the scales again.
  Arms: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of nursing follow-up by phone on the self-efficacy status, pain, and disease activity of individuals with RA using biological agents. The study sample consisted of 64 individuals, including 32 interventions and 32 comparison groups, who met the inclusion criteria. The research was conducted in a randomized controlled experimental study design. In data collection; 'Personal Information Form', 'Arthritis Self-Efficacy Scale', 'Visual Analog Scale' and 'DAS 28' score was used. Descriptive statistics (mean±sd) for numerical variables and frequency distributions for categorical variables were used to evaluate the data.

Individuals in the intervention group participating in the research; 65.6% of them were women and their mean age was 50.12 (±13.200); of the individuals in the comparison group who participated in the study, it was determined that 56.3% of them were female, their mean age was 45.97 (±11.544). There was no difference in self- efficacy, pain, and disease activity in the first evaluation before the nursing follow-up by phone between the individuals in the intervention and comparison group, and as a result of the 24-week nursing follow-up by phone of the individuals in the intervention group after the training, when compared with the individuals in the comparison group who received routine outpatient service; It was noted that there was an increase in self- efficacy, a decrease in pain severity, and a decrease in disease activity.

The self-efficacy, pain, and disease activity of individuals with a diagnosis of RA who use biological agents should be monitored regularly, training needs should be met, telenursing counseling practices should be expanded to increase the effectiveness of education and to manage the process more effectively, and arrangements should be made to enable patients to access telenursing counseling.

DETAILED DESCRIPTION:
The study was conducted in a randomized controlled experimental study design with the aim of determining the effect of nursing follow-up by phone on the self-efficacy status, pain, and disease activity of individuals with RA using biological agents. After the power analysis to calculate the sample size of the study, a total of 64 patients were included in each group with 80% power and 5% margin of error assuming that a minimum difference of 2 points was clinically significant in pairwise comparisons made according to VAS pain scores. In the research, patients who applied nursing follow-up by phone formed the intervention group, and patients who only received routine care formed the control group.

ELIGIBILITY:
Inclusion Criteria:

Having been diagnosed with rheumatoid arthritis for at least 1 year,

* To have received at least 3 doses of biologic agent subcutaneously within the DMARD combination treatment option,
* Not having problems in communicating,
* Having no mental problems, hearing and vision problems,
* Being 18 years or older,
* Being conscious,
* Being able to communicate by phone,
* Applying to Sivas Numune Hospital Rheumatology Polyclinic,
* No planned training by health professionals on RA and biological agent therapy before,
* Agree to participate in the study.

Exclusion Criteria:

Losing one's life during the research period,

* Termination of biological agent treatment for any reason,
* Leaving the research voluntarily.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Arthritis Self-Efficacy Scale | It was administered at the first interview and at 12 and 24 weeks after the completion of the training. Changes from baseline Arthritis Self-Efficacy scores at the end of the 12th and 24th weeks
  It was developed in the United States in 1989 by Lorig et al. to help individuals cope with their arthritis and to measure their self-efficacy perceptions. There are a total of 20 expressions on the 10-digit visual scale, which has 3 sub-scopes: self-efficacy in pain, self-efficacy in functions, and self-efficacy in other symptoms. Turkish validity and reliability study was carried out by Ünsal and Kaşıkçı in 2006.

SECONDARY OUTCOMES:
Pain Visual Analog Scale -VAS | It was administered at the first interview and at 12 and 24 weeks after the completion of the training. Changes from baseline Pain Visual Analog scores at the end of the 12th and 24th weeks
  It is used to convert some values that cannot be expressed through numbers into numeric. Pain experienced by the patient during use in RA; Absence of pain is graded between 0 points and severe pain is scored between 10 points (Gift, 1989).
DAS-28 (Disease Activity Score 28) | It was administered at the first interview and at 12 and 24 weeks after the completion of the training. Changes from baseline DAS-28 (Disease Activity Score 28) scores at the end of the 12th and 24th weeks
  It is a scoring system used to determine rheumatoid arthritis disease activity. The calculation is routinely performed by the physician for all patients by evaluating the number of tender and swollen joints, erythrocyte sedimentation rate, global evaluation of the patient and VAS measurements in a special type calculator. According to the obtained DAS score; DAS 28 ≤2.4 is considered as remission, 2.4-3.6 low disease activity, 3.6-5.5 moderate disease activity, ≥ 5.5 high activity value (Prevoo et al., 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Tel Aydın, Professor, Study Director — Cumhuriyet University
Locations (1):
- Döne Günay, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Gronning K, Lim S, Bratas O. Health status and self-management in patients with inflammatory arthritis-A five-year follow-up study after nurse-led patient education. Nurs Open. 2019 Oct 8;7(1):326-333. doi: 10.1002/nop2.394. eCollection 2020 Jan. PMID 31871717
- [Background] Mollard E, Michaud K. Self-Management of Rheumatoid Arthritis: Mobile Applications. Curr Rheumatol Rep. 2020 Nov 26;23(1):2. doi: 10.1007/s11926-020-00968-7. PMID 33244621
- [Background] Piga M, Cangemi I, Mathieu A, Cauli A. Telemedicine for patients with rheumatic diseases: Systematic review and proposal for research agenda. Semin Arthritis Rheum. 2017 Aug;47(1):121-128. doi: 10.1016/j.semarthrit.2017.03.014. Epub 2017 Mar 22. PMID 28420491
- [Background] Primdahl J, Sorensen J, Horn HC, Petersen R, Horslev-Petersen K. Shared care or nursing consultations as an alternative to rheumatologist follow-up for rheumatoid arthritis outpatients with low disease activity--patient outcomes from a 2-year, randomised controlled trial. Ann Rheum Dis. 2014 Feb;73(2):357-64. doi: 10.1136/annrheumdis-2012-202695. Epub 2013 Feb 5. PMID 23385306
- [Background] Ryan S. Psychological effects of living with rheumatoid arthritis. Nurs Stand. 2014 Dec 2;29(13):52-9. doi: 10.7748/ns.29.13.52.e9484. PMID 25424112
- [Background] Uthman I, Almoallim H, Buckley CD, Masri B, Dahou-Makhloufi C, El Dershaby Y, Sunna N, Raza K, Kumar K, Abu-Saad Huijer H, Tashkandi N, Louw I, Adelowo O. Nurse-led care for the management of rheumatoid arthritis: a review of the global literature and proposed strategies for implementation in Africa and the Middle East. Rheumatol Int. 2021 Mar;41(3):529-542. doi: 10.1007/s00296-020-04682-6. Epub 2020 Aug 26. PMID 32851423
- [Background] Zhang L, Cai P, Zhu W. Depression has an impact on disease activity and health-related quality of life in rheumatoid arthritis: A systematic review and meta-analysis. Int J Rheum Dis. 2020 Mar;23(3):285-293. doi: 10.1111/1756-185X.13774. Epub 2019 Dec 19. PMID 31858731